CLINICAL TRIAL: NCT00464763
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Two-Arm Parallel, Multicenter Study Evaluating the Efficacy and Safety of Dexmedetomidine in the Prevention of Postoperative Delirium in Subjects Undergoing Heart Surgery With Cardiopulmonary Bypass
Brief Title: A Research Study to Evaluate the Effectiveness of Dexmedetomidine in Preventing Delirium After Heart Surgery
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The incidence of post-operative delirium observed from interim blinded data in DEX-06-09 was significantly lower than the current literature in this population.
Sponsor: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DEX-06-06
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2015-11

CONDITIONS: Delirium
Keywords: Mental Health; Neurological Disease; Heart Valve Repair Surgery
MeSH Terms: conditions — Delirium; Psychological Well-Being; Nervous System Diseases | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine (Experimental)
  Interventions: Drug: Dexmedetomidine
- Placebo (PBO) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine
  Arms: Dexmedetomidine
Drug: Placebo
  Arms: Placebo (PBO)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of dexmedetomidine in the prevention of postoperative delirium in subjects undergoing heart valve surgery with or without coronary artery bypass surgery (CABG) using cardiopulmonary bypass (CPB).

DETAILED DESCRIPTION:
Postoperative delirium is an acute decline in cognition and attention which is usually transient but when delirium persists, it can impact cognitive function, morbidity and mortality. Currently, there are no drugs to prevent delirium but dexmedetomidine has the potential to meet this unmet medical need.

Dexmedetomidine is currently approved for use for 24 hours in patients on ventilators in the Intensive Care Unit(ICU). This study is to determine whether or not dexmedetomidine can prevent delirium after heart surgery. Study participation will last from randomization prior to surgery, to 3 days after surgery. Dexmedetomidine will be given through an intravenous catheter beginning at sternal closure and continue throughout the stay in the ICU. Delirium will be assessed prior to surgery and for 72 hours after surgery. This assessment will consist of questions that will evaluate memory and thought process. Thirty days after surgery, questions will be asked regarding the patients feelings about their health status and hospital billing information will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years old) male or female who will undergo elective heart valve surgery (with or without CABG and using CPB) with general anesthesia and require an overnight stay in the ICU following surgery.
* If female, subject is non-lactating and is either:

  1. Not of childbearing potential, defined as post-menopausal for at least 1 year or surgically sterile due to bilateral tubal ligation, bilateral oophorectomy or hysterectomy.
  2. Of childbearing potential but is not pregnant at time of baseline and is practicing one of the following methods of birth control: oral or parenteral contraceptives, doublebarrier method, vasectomized partner, or abstinence from sexual intercourse.
* Subject is American Society of Anesthesiologists (ASA) Physical Status II, III, or IV.
* Subject (or subject's legally authorized representative) has voluntarily signed and dated the informed consent document approved by the Institutional Review Board (IRB).

Exclusion Criteria:

* Cognitive function level by Mini Mental State Exam (MMSE) of ≤ 20 at screening.
* Subject has a positive CAM-ICU result for delirium at Screening.
* Subject requires chronic anti-psychotic therapy.
* Subject has participated in a trial with any experimental drug or experimental implantable device within 30 days prior to the study drug administration, or has ever been enrolled in this study.
* Subject is known to be in liver failure.
* Subject has an anticipated potential for increased intracranial pressure or an uncontrolled seizure disorder or known psychiatric illness that could confound a normal response during study assessment.
* Subject has acute myocardial infarction, HR <50 bpm, SBP <90 mmHg, is hemodynamically unstable requiring systemic inotropic drugs or intra-aortic counterpulsation balloon pump within the last 72 hours.
* Subject is anticipated to require hypothermic circulatory arrest during this surgical procedure.
* Subject has received treatment with a α2-agonist or antagonist (within 14 days of study entry).
* Subject for whom opiates, propofol, Dexmedetomidine or other α2-agonists are contraindicated.
* Subject has, per the investigator's judgment, a known or suspected physical or psychological dependence on an abused drug, other than alcohol.
* Subject has any condition or factor which, in the Investigator's opinion, might increase the risk to the subject.
* Subject is not expected to live more than 60 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-04; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects who experienced any postoperative delirium up to 3 days following surgery | Postoperative period (3-days): Twice daily (6:00 - 9:00 AM and 5:00 - 8:00 PM)
  The presence of postoperative delirium will be determined by the Confusion Assessment Method (CAM-ICU)

SECONDARY OUTCOMES:
Daily percentage of subjects who experienced postoperative delirium | At each day during 3-day postoperative delirium
Duration of postoperative delirium as determined by CAM-ICU up to 3 days post surgery | Up to 3 days post surgery
Postoperative use of all analgesics | During postextubation period (Approximately 3 days)
Time to extubation after arrival in ICU | From the time of ICU arrival to the time of ICU discharge (Approximately 3 days)
Length of ICU stay | From the time of ICU arrival to the time of ICU discharge (Approximately 3 days)

CONTACTS AND LOCATIONS:
Overall Officials: Paula Bokesch, MD, Study Director — Hospira, now a wholly owned subsidiary of Pfizer
Locations (11):
- United States (11):
  - Loma Linda University, Loma Linda, California
  - Midatlantic Cardiovascular Associates, Towson, Maryland
  - Genesys Cardiovascular and Thoracic Surgical Associates, Grand Blanc, Michigan
  - Cooper University Hospital, Camden, New Jersey
  - Cleveland Clinic, Cleveland, Ohio
  - Cardiothoracic and Vascular Surgical Specialists, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas
  - Texas Heart Institute, Houston, Texas
  - University of Virginia Health System, Dept. of Anesthesiology, Charlottesville, Virginia
  - Santara Norfolk General Hospital, Norfolf, Virginia